CLINICAL TRIAL: NCT04086134
Title: The FruGut Study: Physiological, Microbiological and Metabolomic Effects of Fruit Products
Brief Title: Physiological, Microbiological and Metabolomic Effects of Fruit Products
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Queen Mary University of London (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HR-17/18-7858
Record Dates: First submitted 2019-06-20; First posted 2019-09-11 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Constipation - Functional
Keywords: constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention fruit products 1 (Experimental): Three servings of fruit products per day for 4 weeks.
  Interventions: Other: Fruit Products
- Intervention fruit products 2 (Experimental): Three servings of fruit products per day for 4 weeks.
  Interventions: Other: Fruit Products
- Control fruit products (Placebo Comparator): Three servings of control fruit products per day for 4 weeks.
  Interventions: Other: Fruit Products

INTERVENTIONS:
Other: Fruit Products — Fruit Products with the potential to improve constipation-related outcomes

SUMMARY:
This study is a randomised, parallel group, controlled trial, comparing the effects of fruit products as to their physiological, microbiologic and metabolomic effects on the gut, as well as their effects on the dietary intake and quality in healthy people with constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65 years.
2. Individuals meeting the Rome IV criteria for functional constipation, in addition to having <7 bowel movements per week and hard or lumpy stools present in ⩾25% of their defecations (defined as Type 1 & 2 of the Bristol Stool Form Scale).
3. Individuals who are willing to consume fruit products for 4 weeks.
4. Individuals who consume <30g of fibre per day
5. Individuals with a BMI of 18.5-29.99 kg/m2.
6. Individuals able to give informed consent.

Exclusion Criteria:

1. Females who report to be pregnant or lactating.
2. Regular consumers of the fruit products used in the intervention arm 1 (3 or more portions per week).
3. Allergy, intolerance or dislike of the fruit products used in this intervention.
4. Sulphite allergy or sensitivity.
5. Ongoing alcohol, drug or medication abuse.
6. Major medical condition (diabetes, psychiatric or current eating disorders), gastrointestinal disease (e.g. inflammatory bowel disease, coeliac disease) or history of previous GI surgery, except cholecystectomy, appendicectomy and haemorrhoidectomy.
7. Medications which affect their gut physiology, function and symptoms in the last 4 weeks, and individuals who are not willing or cannot discontinue them.
8. Frequent use of rescue laxatives.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in faecal weight between baseline and week 4 | week 4
  Change in 7-day faecal weight

SECONDARY OUTCOMES:
Faecal microbiome diversity | week 0 and 4
  Global microbiota composition (α-diversity, β-diversity)
Faecal microbiome | week 0 and 4
  Ιndividual phyla, family, genera, species and strains of the faecal gut microbiome (absolute and change).
Faecal metabolomic profile | week 0 and 4
  Faecal metabolomic profile (absolute and change) measured using proton nuclear magnetic resonance
Urine metabolomic profile | week 0 and 4
  Urine metabolomic profile (absolute and change) measured using proton nuclear magnetic resonance
Faecal short-chain fatty acids | week 0 and 4
  Faecal short-chain fatty acids concentration (absolute and change)
Faecal water content | week 0 and 4
  Faecal water content (absolute and change) measured through lyophilisation
Faecal pH | week 0 and 4
  Faecal pH (absolute and change)
Stool output | week 0 and 4
  Assessed using 7-day diaries and the Bristol Stool Form Scale (absolute and change)..
Individual gastrointestinal symptoms | week 0 and 4
  The 7-day diaries contain a short questionnaire for each bowel movement to monitor completeness, spontaneity, straining and need for manual maneuvers. The validated Gastrointestinal Symptom Rating Scale will be used over a 7-day period
Gastrointestinal symptoms - PAC-SYM | week 0 and 4
  The validated questionnaire Patient Assessment of Constipation Symptoms (PAC-SYM) will be used (absolute and change).
Gastrointestinal symptom severity questionnaire - CCCS | week 0 and 4
  The validated questionnaire Cleveland Clinic Constipation Score (CCCS) will be used (absolute and change).
Dietary intake | week 0 and 4
  Dietary intake (absolute and change) will be recorded in 7-day food and drink diaries
Constipation-related quality of life | week 0 and 4
  Constipation-related quality of life (absolute and change) which will be measured with the condition-specific validated Patient Assessment of Constipation Quality of Life (PAC-Qol) questionnaire. PAC-QoL is a self-report 28-item tool that uses a 5-point Likert scale ranging from "Not at all" to "Extremely".
Whole and regional gut transit time/pH | week 0 and 4
  Whole gut transit time and regional gut pH (absolute and change) will be assessed in a subset of participants (n=39), by using a motility capsule (SmartPill ®, Medtronic)
Acceptability of interventions | week 0 and 4
  Acceptability of the interventions measured using a questionnaire that included 3- and 4-point likert scales and open-text answers
Compliance | week 0 and 4
  Compliance to the study interventions will be measured using specific questions relevant to the intervention received in the food and drink diary completed at week 4, by regular phone calls with participants throughout the intervention period, and by the number of unconsumed fruit products returned by the participants after the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Whelan, MSc, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No